CLINICAL TRIAL: NCT03607045
Title: Headless Screws Versus Bouquet in Intramedullar Fixation of Boxer's Fracture: A Randomized Clinical Trial
Brief Title: Headless Screws x Bouquet in Boxer's Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculdade de Medicina do ABC (Other)
Responsible Party: Principal Investigator, Marcio Aurelio Aita, Affiliated Professor, Faculdade de Medicina do ABC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 311718
Record Dates: First submitted 2018-04-30; First posted 2018-07-31 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Boxer's Fracture
Keywords: Boxer's Fracture

STUDY DESIGN:
Intervention Model Description: two groups homogeneous
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Placebo Comparator): bouquet technique
  Interventions: Device: headless screw
- test group (Active Comparator): headless screw
  Interventions: Device: headless screw

INTERVENTIONS:
Device: headless screw — headless screw group

SUMMARY:
Despite the high prevalence (20% of the hand fractures) of unstable neck metacarpals fractures (boxer's fractures) there is still no consensus concerning the preferred method and ideal moment of treatment, especially in active patients where the time or type of management can have a strong psychological impact on the outcomes.

The use of intramedullar technique (headless intramedular screws or bouquet technique fixation) as definitive treatment of unstable boxer's fractures in active patients at the first week, may be a good choice of treatment. This technique is fast, safe, minimally invasive and easily performed reproducible method, without address the extensor tendon to prevent tendon adhesion and joint stiffness, unable earlier functional recovery and shorten the working return time of these patients. Choose a reproducible and effective method, which presents a cost / benefit compatible with our reality.

The goal of the present study is to compare working return time, VAS (visual analogue score), quick DASH (disability arm, shoulder and hand) and radiographic outcomes of two methods of definitive internal fixation in active patients in boxer's fractures, operated in the first week.

DETAILED DESCRIPTION:
A double center, parallel group, prospective, randomized clinical trial was conducted at the department of Hand Surgery, ABC University hospital, Santo Andre, Brazil and Hospital Mãe de Deus, Porto Alegre, Brazil. Two implants used for fixation in closed reduction of boxer's fractures were compared: the headless cannulated screws (Synthes®, Davos) and the Bouquet technique with k-wires (Synthes®, Davos). The protocol was approved by the local research ethics committee. All patients received, signed and are aware of what was recommended in the Informed Consent (IC). Inclusion criteria were; presence of an acute (0 to 7 days), closed and simple fracture of the metacarpal neck, absence of an ipsilateral injury or deformity, Start January 2017.

ELIGIBILITY:
Inclusion Criteria:

* presence of an acute (0 to 7 days), closed and simple fracture of the metacarpal neck, absence of an ipsilateral injury or deformity, presence of an angulation of over 40 degrees in oblique plane imaging, being 18 years of age or older, having acquired a master's degree or still being a student, and being an employee in a social-professional environment with mild physical activities.

Exclusion Criteria:

* elderly, children, mental ness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
patient outcome reported | 6 months
  QuickDASH

CONTACTS AND LOCATIONS:
Overall Officials: Marcio Aurelio a Aita, Principal Investigator — Centro Universitário FMABC
Locations (1):
- Marcio Aurelio Aita, São Bernardo do Campo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided